CLINICAL TRIAL: NCT04437186
Title: The Effectiveness of a Recovery Program for People With Mental Illness: A Multicenter Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B-BR-108-064
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-01

CONDITIONS: Mental Illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery group (Experimental): The recovery program has 2 phases and consists of 20 classes, 1.5 hour per class and one class per week. We will introduce concepts of recovery and personal strengths in phase 1. Then, we will help participants to set goals and implement their plans in phase 2. Participants will fill out all questionnaires during the recruitment meeting.They will fill out the same questionnaires plus the course satisfaction survey in the end of phase 1 and 2. Six months later, participants will receive a follow-up interview and fill out the questionnaires again.
  Interventions: Behavioral: Recovery program
- Control group (No Intervention): The control group will receive a spiritual book and complete the questionnaires at the same time as the recovery group.

INTERVENTIONS:
Behavioral: Recovery program — The researchers designed a recovery group suited to Taiwanese with mental illness, according to content of the Pathways to Recovery (PTR): A Strengths Recovery Self-Help Workbook (Ridgway et al., 2002) and recovery-related literature (Davidson et al., 2005; Ridgway, 2001)
  Arms: Recovery group

SUMMARY:
Recovery-oriented approach has been the main trend in mental health field. However, few recovery-oriented programs are available in Taiwan, and many Taiwanese people with mental illness don't understand the concepts of recovery. A program which provides recovery knowledge and assists in setting recovery goals is beneficial for Taiwanese people with mental illness. Hence, this study aimed to investigate the effectiveness of a recovery program for people with mental illness.

DETAILED DESCRIPTION:
This is a randomized control trial. Participants will be recruited from the psychiatric rehabilitation organizations in Taiwan. They will be randomly assigned to the intervention group or control group. The recovery program has 2 phases and consists of 20 classes, 1.5 hour per class and one class per week. We will introduce concepts of recovery and personal strengths in phase 1. Then, we will help participants to set goals and implement their plans in phase 2. Participants will fill out five questionnaires during the recruitment meeting, including Stages of Recovery Scale, Medical Outcomes Study Social Support Survey, The Hope Scale, Rosenberg Self-Esteem Scale and Brief Symptom Rating Scale-50. They will fill out the same questionnaires plus the course satisfaction survey in the end of phase 1 and 2. Six months later, participants will receive a follow-up interview and fill out the questionnaires again. The control group will receive a spiritual book and complete the questionnaires at the same time as the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mental illness
* lived in community

Exclusion Criteria:

-

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Stages of Recovery Scale (SRS) | Change from Baseline at 10 weeks, 20 weeks and 44 weeks
  The scale consists of 45 items, with six subscales: the sense of hope, disability management/taking responsibility, regaining autonomy, social functioning/role performance, overall well-being, and willingness to help. It has good internal consistency and proper construct validity. The SRS utilizes a 4-point rating scale: never (0), seldom (1), sometimes (2), and often (3). Higher scores indicate better recovery. The developers also provide the cutoff scores for four recovery stages: Stage 1 (overwhelmed by the disability), 0-57; Stage 2 (struggling with disability), 58-90; Stage 3 (living with disability), 91-119; and Stage 4 (living beyond disability), 120-135.

SECONDARY OUTCOMES:
Medical Outcomes Study Social Support Survey (MOS-SS) | Change from Baseline at 10 weeks, 20 weeks and 44 weeks
  The Medical Outcomes Study Social Support Survey (MOS-SS) is a multidimensional, self-administered instrument that addresses all five functions of an interpersonal relationship to assess the various functional dimensions of social support, including emotional , informational, tangible, affectionate, and positive interaction (Sherbourne & Stewart, 1991).For each item, the respondents were asked to indicate how often each support was available to them if they needed it. Response options were none of the time (1), a little of the time (2), some of the time (3), most of the time (4), and all of the time (5). For each scale, simple algebraic sums were computed, and then the raw scale scores were transformed into a scale of 0 to 100. The higher the score, the better the perception of social support. The reliability and validity of the measure in an American population of adults with chronic illness have been established (Sherbourne & Stewart, 1991).
The Hope Scale (THS) | Change from Baseline at 10 weeks, 20 weeks and 44 weeks
  The THS is a self-report measure based on the principle that hope is a cognitive set based on an individual's agency (a sense of successful determination in being able to achieve one's goals and a perceived efficacy for initiating and sustaining action toward goal attainment) and pathways (an individual's cognitive appraisal of his or her ability to overcome obstacles and achieve these goals) (Synder et al., 1991). The measure includes 12 items, four measuring pathways and four measuring agency, and four "filler" items that are not used for scoring. The measure yields scores for the agency and pathways subscales, as well as a total score. Across a number of different samples, alphas ranged from .64 to .80 for the pathways subscale, .71 to .77 for the agency subscale, and from .74 to .84 for the total score (Snyder et al., 1997).
Rosenberg Self-Esteem Scale (RSE) | Change from Baseline at 10 weeks, 20 weeks and 44 weeks
  The purpose of the 10 item RSE scale is to measure self-esteem. As the RSE is a Guttman scale, scoring can be a little complicated. Scoring involves a method of combined ratings. Low self-esteem responses are "disagree" or "strongly disagree" on items 1, 3, 4, 7, 10, and "strongly agree" or "agree" on items 2, 5, 6, 8, 9. Two or three out of three correct responses to items 3, 7, and 9 are scored as one item. One or two out of two correct responses for items 4 and 5 are considered as a single item; items 1,8, and 10 are scored as individual items; and combined correct responses (one or two out of two) to items 2 and 6 are considered to be a single item. The scale can also be scored by totalling the individual 4 point items after reverse-scoring the negatively worded items.
Brief Symptom Rating Scale-50 (BSRS-50) | Change from Baseline at 10 weeks, 20 weeks and 44 weeks
  The BSRS comprises 50 items, which best reflect the original ten symptom dimensions and three indices of psychopathology from the SCL-90-R.
  It is self-rated by individuals on a 5-point scale of symptom severity distress (0-4). It can measure nine primary and one additional symptom dimension of psycho-pathology, as well as there indices of distress- General Severity Index (GSI), Positive Symptom Distress Index (PSDI), and Total Number of Positive Symptoms (PST).

OTHER OUTCOMES:
Qualitative data | At 10 weeks, 20 weeks and 44 weeks
  The course discussion of the end of phase 1 and phase 2 will be recorded. In addition, the participants of the intervention group will be interviewed at follow up. Those qualitative data will be transcribed and analyzed.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan